CLINICAL TRIAL: NCT00787462
Title: Evaluation of Pregabalin in Idiopathic Small Fiber Neuropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Restrictive inclusion criteria/limited pool of suitable subjects with SFN.
Sponsor: University of Alberta (Other)
Collaborators: Capital Health, Canada (Other)
Responsible Party: Principal Investigator, Zaeem Siddiqi, Associate Professor, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ZAS-2007-HC-01
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2010-09

CONDITIONS: Small-Fiber Neuropathy
Keywords: Neuropathic; Neuropathic pain; Nerve pain; Pain; Chronic pain; Pregabalin; Lyrica; Small fiber neuropathy; Neuropathy
MeSH Terms: conditions — Small Fiber Neuropathy; Neuralgia; Pain; Chronic Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Available as 75 mg capsules. Subjects will begin Phase 1 treatment on either pregabalin (or placebo) 75mg BID (1 capsule BID) for one week then increasing to 150mg BID or placebo (2 capsules BID) for a further 7 weeks. During this period patients will be allowed to taper the drug to 225mg a day (75mg in am, 150mg in pm) or (75mg BID) if they develop significant adverse effects on the higher dose. After 8 weeks Phase 1 treatment subjects will taper study medication to 75mg BID or placebo (1 capsule BID) for 7 days and then continue taking placebo (1 capsule) for 7 additional days prior to the crossover. After the taper and washout, Phase 2 will begin using the alternate treatment and will follow the same dosing regime as Phase 1 for the remaining 10 weeks.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Available as 75 mg capsules. Subjects will begin Phase 1 treatment on either pregabalin (or placebo) 75mg BID (1 capsule BID) for one week then increasing to 150mg BID or placebo (2 capsules BID) for a further 7 weeks. During this period patients will be allowed to taper the drug to 225mg a day (75mg in am, 150mg in pm) or (75mg BID) if they develop significant adverse effects on the higher dose. After 8 weeks Phase 1 treatment subjects will taper study medication to 75mg BID or placebo (1 capsule BID) for 7 days and then continue taking placebo (1 capsule) for 7 additional days prior to the crossover. After the taper and washout, Phase 2 will begin using the alternate treatment and will follow the same dosing regime as Phase 1 for the remaining 10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Available as 75 mg capsules. Subjects will begin Phase 1 treatment on either pregabalin (or placebo) 75mg BID (1 capsule BID) for one week then increasing to 150mg BID or placebo (2 capsules BID) for a further 7 weeks. During this period patients will be allowed to taper the drug to 225mg a day (75mg in am, 150mg in pm) or (75mg BID) if they develop significant adverse effects on the higher dose. After 8 weeks Phase 1 treatment subjects will taper study medication to 75mg BID or placebo (1 capsule BID) for 7 days and then continue taking placebo (1 capsule) for 7 additional days prior to the crossover. After the taper and washout, Phase 2 will begin using the alternate treatment and will follow the same dosing regime as Phase 1 for the remaining 10 weeks.
  Other Names: Lyrica
  Arms: Active
Drug: Placebo — Available as 75 mg capsules. Subjects will begin Phase 1 treatment on either pregabalin (or placebo) 75mg BID (1 capsule BID) for one week then increasing to 150mg BID or placebo (2 capsules BID) for a further 7 weeks. During this period patients will be allowed to taper the drug to 225mg a day (75mg in am, 150mg in pm) or (75mg BID) if they develop significant adverse effects on the higher dose. After 8 weeks Phase 1 treatment subjects will taper study medication to 75mg BID or placebo (1 capsule BID) for 7 days and then continue taking placebo (1 capsule) for 7 additional days prior to the crossover. After the taper and washout, Phase 2 will begin using the alternate treatment and will follow the same dosing regime as Phase 1 for the remaining 10 weeks.
  Other Names: Visually Identical Placebo
  Arms: Placebo

SUMMARY:
Idiopathic Small Fiber Neuropathy (called SFN for short), is a condition where nerves that sense pain have become damaged, and often painful. SFN pain is common, and it can affect sleep, memory, health and overall quality of life.

Pregabalin is a drug commonly used to treat painful conditions, like nerve pain. It has been available to doctors for many years, and many studies have been performed to evaluate its effectiveness. In these studies, pregabalin has been shown to be very effective in the treatment of nerve pain, with fewer side effects than many other medications currently available. The purpose of the study is to determine if pregabalin relieves pain more effectively than a pill containing no medication (called a placebo). The study will also investigate any side effects as well as the effectiveness and safety of the medication.

DETAILED DESCRIPTION:
Painful small fiber sensory neuropathy (SFN) is relatively common and a disabling medical condition. It is the most common type of painful sensory neuropathy in patients older than 50 years of age. It is defined as a neuropathy that exclusively or predominantly affects the A-δ (small myelinated) and nociceptive C (unmyelinated) nerve fibers and their functions. The neuropathic pain associated with SFN is described by the patients as burning ("feet are on fire"), sharp ("knife-like, jabbing or pins and needles"), shooting, and aching pain in the toes and feet. The feet are described as tingling, numb, or feeling tight, wooden or dead. The pain is disabling and often exacerbated at night interfering and disrupting the sleep pattern. Allodynia and cramps may also occur. Some patients also describe pressure induced pain in their feet with standing and walking. The autonomic nerves may be involved leading to increased or decreased sweating, facial flushing, skin discoloration and erectile dysfunction in up to 40% of males. On examination there is a dramatic mismatch between the symptoms and observable deficits in SFN. Only abnormal findings are the loss of pinprick and temperature sensations in feet that may extend up to the knees. Touch sensation may be diminished but other sensations are usually preserved. By definition, patients with SFN are allowed to have minor involvement of large fibers distally with reduced vibration in toes but the ankle reflexes are usually preserved.

This study will be of a crossover design thus minimizing the number of subjects needed. Each patient will act as his/her own control. Previous studies of pregabalin have shown that the desired effect is achieved by eight weeks of treatment. Therefore each patient will start on either placebo or pregabalin. They will be assessed on this treatment arm for eight weeks. There will be a two-week drug tapering and washout period before switching treatments, followed by re-assessment for an additional eight weeks. This design minimizes the amount of time that the patient will be treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic SFN (based on clinical and electrodiagnostic criteria).
* Each day for 7 days prior to Visit 2 (Washout) they must complete a modified Quadruple Visual Analogue Scale₁ showing moderate to severe pain (i.e. a daily mean rating score of ≥ 4).
* As the safety of pregabalin in pregnancy has not been established, females of childbearing potential must have a negative βHCG serum and agree to practice acceptable birth control methods.
* All subjects must have screening laboratory values that are within normal limits or abnormal values that are deemed not clinically significant by the Principle Investigator.

Exclusion Criteria:

* Have a psychological or psychiatric condition that may hinder their ability to provide important information
* History of psychosis, drug or alcohol abuse history within the last year
* Malignancy within the last 2 years (except skin cancer)
* Clinically significant conditions (including but not limited to cardiovascular or hepatic diseases), and seizure disorders.
* Subjects with an abnormal 2-hour glucose tolerance test (i.e., glucose >7.8 mmol/l) will be excluded under "clinically significant conditions" as stated above.
* May not have participated in a previous trial of pregabalin, have a history of intolerance or hypersensitivity to pregabalin.
* Patients with renal impairment (CrCl < 60 ml/min) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Neuropathic pain score | 21 weeks
  Measured difference in the mean neuropathic pain score recorded in daily pain assessment scores between the pregabalin treatment phase (escalating twice daily dose of 75mg, 150mg) versus placebo treatment phase.

SECONDARY OUTCOMES:
Quality of life measures | 21
  Measure differences in the mean scores of other quality of life measures between the pregabalin treatment phase (escalating twice daily dose of 75mg, 150mg) versus placebo treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Zaeem A Siddiqi, MD, PhD, Principal Investigator — MD, Profesor of Medicine, Neurology
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to insufficient recruitment.